CLINICAL TRIAL: NCT00625924
Title: Sensory Morbidity Following Breast Surgery
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-009
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Breast Cancer
Keywords: Plastic surgery; reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- 1: autogenous tissue breast reconstruction
  Interventions: Behavioral: questionnaires
- 2: tissue expander/implant breast reconstruction
  Interventions: Behavioral: questionnaires
- 3: mastectomy alone
  Interventions: Behavioral: questionnaires

INTERVENTIONS:
Behavioral: questionnaires — Patients will be evaluated at one time point using the Breast Sensation Assessment Score (BSAS©), the SF-36 Health Survey, the MSKCC BREAST Q, the Brief Pain Inventory, the Hopwood Body Image Scale, the Profile of Mood States - Brief Version (POMS - BRF), and the 'Patient Demographic and Treatment Information Form'
  Groups: 1
Behavioral: questionnaires — Patients will be evaluated at one time point using the Breast Sensation Assessment Score (BSAS©), the SF-36 Health Survey, the MSKCC BREAST Q, the Brief Pain Inventory, the Hopwood Body Image Scale, the Profile of Mood States -Brief Version (POMS - BRF), and the 'Patient Demographic and Treatment Information Form'
  Groups: 2
Behavioral: questionnaires — Patients will be evaluated at one time point using the Breast Sensation Assessment Score (BSAS©), the SF-36 Health Survey, the MSKCC BREAST Q, the Brief Pain Inventory, the Hopwood Body Image Scale, the Profile of Mood States -Brief Version (POMS - BRF), and the 'Patient Demographic and Treatment Information Form'
  Groups: 3

SUMMARY:
The goal of the study is measure breast sensations after breast surgery. The results of this study will help surgeons better understand breast sensations and may improve the way surgery is done.

ELIGIBILITY:
Inclusion Criteria:

* The Samples used will be derived from three cohorts below and will only include patients who have completed mastectomy or reconstruction within 1-5 years of enrollment.
* Patients who have undergone immediate, two-stage expander/implant postmastectomy reconstruction
* Patients who have undergone immediate, autogenous tissue flap reconstruction following mastectomy
* Patients who have undergone mastectomy alone
* Patients at least 21 years of age
* Patients who completed mastectomy ± immediate post-mastectomy reconstruction at least one year but no longer than five years prior to study entry

Exclusion Criteria:

* Patients who have had any of the following:
* delayed reconstruction (no reconstruction at time of surgery) combined autogenous tissue/implant breast reconstruction, and/or
* Patients who have a pre-surgical history of complex regional pain syndrome
* Patients who have had radiation therapy
* Patients who have had a local recurrence
* Patients who do not speak the English language (validated translations of key questionnaires are not available).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2008-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the prevalence, severity and level of distress of subjective breast sensations following mastectomy and postmastectomy reconstruction. | conclusion of the study

SECONDARY OUTCOMES:
To compare sensory morbidity following three types of breast surgery: tissue expander/implant breast reconstruction, autogenous tissue reconstruction, and no reconstruction. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pusic, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org